CLINICAL TRIAL: NCT00095186
Title: A Multi-Center, Phase 2, Open Label Study of Safety and Efficacy of Oral Recombinant Human Lactoferrin (rhLF) Monotherapy in Patients With Advanced Renal Cell Carcinoma (RCC), Who Have Failed at Least One Regimen of Systemic Therapy for RCC
Brief Title: Safety/Efficacy Study of Oral Recombinant Human Lactoferrin in Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Agennix (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LF-0209; NCT00099034 (obsolete NCT alias)
Record Dates: First submitted 2004-11-01; First posted 2004-11-02 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-04

CONDITIONS: Carcinoma, Renal Cell
Keywords: Cancer; Metastatic; Kidney; Refractive; Lactoferrin; Oral
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms; Neoplasm Metastasis

INTERVENTIONS:
Drug: Recombinant Human Lactoferrin

SUMMARY:
The purpose of this study is to determine if orally-administered recombinant human lactoferrin is effective in the treatment of advanced renal cell carcinoma (RCC) in patients who have failed at least one prior systemic therapy for RCC.

DETAILED DESCRIPTION:
This is an open label, multi-center Phase 2 study. Approximately 40 patients will be enrolled in a single study arm. RhLF, at a dose of 1.5 g [1 vial], twice a day (b.i.d.), will be administered orally for two cycles each of 12 consecutive weeks followed by 2 weeks off. A maximum of two additional cycles may be given if an objective response is obtained or if the patient has stable disease and no increase in the size of the target tumor(s) relative to either the Screening CT or the most recent CT measurement, measured according to RECIST prior to the additional cycle(s). Response and progression-free survival will be evaluated for the first 20 patients enrolled. If no patient has an objective response and less than 10% of the patients are alive and progression-free at 14 weeks from the start of Study Drug, then the study will be terminated. If in either Cycle 3 or Cycle 4, more than three out of the first ten patients or more than six out of the first twenty patients entering the cycle experience a Grade 3 or 4 Study-Drug-related adverse event, no further patients will advance into Cycle 3 or Cycle 4.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically confirmed, advanced or metastatic RCC with predominantly clear cell histology that is unresectable or medically inoperable.
* Experienced and failed at least one regimen of systemic therapy for RCC with CT documentation of disease progression.
* A previous CT (4 weeks or more prior to the Screening CT) showing progression of the target tumor(s) compared to a prior CT no more than 9 months previously
* At least one target tumor lesion is measurable at Screening with CT scan, according to RECIST, and not previously irradiated
* Karnofsky performance status of ≥70 (ECOG <2)
* Able to understand and sign an informed consent

Exclusion Criteria:

* Significant sarcomatoid, spindle cell, or nuclear grade 4 histology
* Significant non-clear cell RCC (for example, papillary, chromophobe, collecting duct, granular, or unclassified RCC)
* Total bilirubin >1.5 mg/dL
* Serum creatinine >2.0 mg/dL
* Hemoglobin <10.0 g/dL
* Absolute neutrophil count <2000/mm3
* Lymphocytes <800/mm3
* Platelet count <100,000/mm3
* AST (SGOT) or ALT (SGPT) ≥2.5 x institutional upper limit of normal
* Serum calcium >11.5 mg/dl
* International Normalized Ratio of Prothrombin Time (INR) >1.2
* FEV1 <60% predicted or FVC <60% predicted by spirometry (both are to be measured)
* Existing or history of brain metastases
* History of allergic reactions to compounds of similar chemical or biologic composition to the Study Agent rhLF
* Active ischemic heart disease, symptomatic congestive heart failure
* Serious active infection
* Psychiatric illness/social situations that would limit compliance with study requirements
* Autoimmune diseases (e.g., systemic lupus erythematosus, multiple sclerosis or ankylosing spondylitis)
* Other malignancies, except non-melanoma skin cancer, within 5 years of study entry
* Radiotherapy within 4 weeks prior to study treatment start
* Corticosteroid therapy within 4 weeks prior to treatment start, with the exception of inhaled or topical steroids
* Chemotherapy/Immunotherapy (e.g., IL-2, INFα, tumor vaccine) within 4 weeks prior to study treatment start
* Known HIV positive
* Receipt of any investigational medication within 30 days prior to participation in the study
* Pregnant or lactating patients, or fertile female patients with a positive pregnancy test (serum β-human chorionic gonadotropin [β-HCG] at Screening and on Day 1 prior to the first dose), or fertile female patients unwilling to use adequate contraception prior to study entry, during treatment and 30 days after completion of treatment
* Sexually active male patients unwilling to practice contraception while participating on this study and up to 30 days after completion of treatment
* Unable to take liquid medication by mouth or feeding tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-09; Study Completion 2007-03

PRIMARY OUTCOMES:
Best Overall Response rate using RECIST criteria
14-WeekProgression-Free Survival (PFS) rate

SECONDARY OUTCOMES:
4 month and 8 month Progression-Free Survival (PFS) rates
Median progression-free survival
Median Overall Survival (OS) and 1-year OS rate
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Ernest W. Yankee, Ph.D., Study Chair — Agennix, Inc.
Locations (6):
- United States (6):
  - University of California, Los Angeles, California
  - Stanford University School of Medicine, Stanford, California
  - The University of Chicago Medical Center, Chicago, Illinois
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - M.D. Anderson Cancer Center, Houston, Texas
  - VA Medical Center/Baylor College of Medicine, Houston, Texas

REFERENCES:
- See also: Sponsor's Home Web Page — http://www.agennix.com